CLINICAL TRIAL: NCT06133348
Title: Promoting Resilience in Women With Breast Cancer
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gabrielle Rocque, Associate Professor of Medicine, Division of Hematology & Oncology; Division of Gerontology, Geriatrics, & Palliative Care, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 300011028; 2027123 (Other Grant/Funding Number: Daiichi Sankyo)
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRISM Intervention (Experimental): This single-arm pilot study will (1) test feasibility, acceptability, and appropriateness of the PRISM intervention in individuals with breast cancer, (2) elicit patient perspectives on elements for future adaptation or expansion to meet the unique needs of women with breast cancer, (3) assess trajectory of patient-reported outcomes and biological measures of stress for patients with breast cancer receiving the PRISM intervention.
  Interventions: Behavioral: Promoting Resilience in Stress Management Intervention

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management Intervention — PRISM is a manualized, brief, skills-based intervention targeting four resilience resources; PRISM is delivered by trained intervention staff (called "coaches" within the PRISM program). Session 1, Stress-Management. Session 2, Goal setting. Session 3, Cognitive Restructuring. Session 4, Meaning-Making. Session 5 (optional), Coming Together. Session 6 (optional) involved advance care planning to discuss.

SUMMARY:
The PRISM (Promoting Resilience in Stress Management) intervention is an evidence-based program that builds resilience. This program was developed in adolescent and young adult oncology and utilizes centrally administered skills-based coaching to bolster positive psychological tools known as resilience resources. These resources include stress management, goal-setting, and positive reframing. Previous studies using this intervention have found PRISM to be successfully administered remotely and it has improved resilience, psychological distress, hope, and quality of life. Among adult caregivers, PRISM has shown to improve resilience, self-efficacy, and engagement with medical care. While PRISM successfully targets distress and associated downstream consequences known to be experienced by breast cancer survivors, it has not been utilized in adults with cancer or in marginalized communities. Adapting this intervention to this context will require the testing of the intervention and, importantly, tailoring to meet the needs of women with breast cancer, particularly those of marginalized populations who may uniquely benefit from this intervention.

DETAILED DESCRIPTION:
This single-arm pilot study will (1) test feasibility, acceptability, and appropriateness of the PRISM intervention in individuals with breast cancer, (2) elicit patient perspectives on elements for future adaptation or expansion to meet the unique needs of women with breast cancer, (3) assess trajectory of patient-reported outcomes and biological measures of stress for patients with breast cancer receiving the PRISM intervention.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing neoadjuvant chemotherapy with early-stage breast cancer, women undergoing treatment for metastatic breast cancer

Exclusion Criteria:

* patients who do not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 43 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Rocque, MD, MSPH, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRISM Intervention
Started | 43
Completed | 33
Not Completed | 10
Not completed — Death | 3
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 43
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 55 [44 to 61]
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 17
  More than one race | 1
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Education [Count of Participants; unit: Participants] — Highest level of education obtained at the start of the intervention
  Participants
    High School, No Degree | 2
    High School Graduate/GED | 5
    Some College | 12
    Associate's Degree | 8
    Bachelor's Degree | 5
    Advanced Degree | 11
Martial Status [Count of Participants; unit: Participants]
  Single, Never Married | 5
  Married/Partnered | 18
  Separated/Divorced | 18
  Widowed | 2
Employment Status [Count of Participants; unit: Participants] — Employment status at the start of the intervention
  Participants
    Not Employed | 17
    Part-time | 6
    Full-time | 13
    Retired | 7
Insurance Coverage [Count of Participants; unit: Participants] — Insurance coverage at the start of the intervention
  Participants
    Private | 21
    Medicaid | 10
    Medicare | 9
    Medicaid/Medicare Dual Enrollment | 1
    Veterans Administration/Military | 1
    Other | 1
Rurality [Count of Participants; unit: Participants] — Rurality is derived from Rural-Urban Commuting Area (RUCA) codes created using the participant's place of residence
  Participants
    Rural | 2
    Urban | 40
    Unknown | 1
Area Deprivation Index [Count of Participants; unit: Participants] — More deprived neighborhoods are link to worse health outcomes when compared to those in neighborhoods that are less deprived. Index is based on the participant's place of residence.
  Participants
    Least Deprived | 31
    Most Deprived | 10
    Unknown | 2
Cancer Therapy Type [Count of Participants; unit: Participants]
  Neoadjuvant | 21
  Adjuvant | 11
  Metastatic | 11
Cancer Stage [Count of Participants; unit: Participants] — Cancer stage was captured from the participant's electronic medical record which utilizes the American Joint Committee on Cancer (AJCC) TNM system. The TNM system take into account tumor size, if cancer has spread to lymph nodes, and metastasis to distant organs. Stage numbers often represent the degree to which cancer has spread. A lower stage number indicates a more early-stage cancer that generally has a good prognosis. As the stage number increases, the cancer becomes more advanced and more difficult to treat.
  Participants
    Stage I | 2
    Stage II | 28
    Stage III | 3
    Stage IV - New Diagnosis | 5
    Stage IV - Recurrent Diagnosis | 5
Cancer Subtype [Count of Participants; unit: Participants] — HR is hormone receptor and can be positive or negative. HR+ indicates that tumor cells have receptors for estrogen and progesterone that promotes tumor growth. HR- indicates that tumor cells do not have hormone receptors. HER2 is human epidermal growth factor receptor 2 and can be positive of negative. HER2+ indicates that tumor cells have higher levels of HER2/neu and is associate with more aggressive breast cancers.
  Participants
    HR+HER2+ | 12
    HR+HER2- | 20
    HR-HER2+ | 2
    HR-HER2- | 7
    HR+HER2 unknown | 1
    HR-HER2 unknown | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Only females were recruited.
  Participants
    Female | 43
    Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of PRISM
Description: Feasibility was defined as 70% of participants completing all sessions and pre/post surveys.
Time Frame: 8 months 4 weeks
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 43
Participants
  Completed both pre-post surveys and all 6 sessions | 33
  Didn't complete PRISM | 10

2. Secondary Outcome: Acceptable, Appropriate, and Feasible
Description: Acceptability, appropriateness, and feasibility of the intervention were measured using the Acceptability of Intervention Measure (AIM; scored 1-5), Intervention Appropriateness Measure (IAM; scored 1-5), and Feasibility of Intervention Measure (FIM; scored 1-5). Higher scores indicated better outcomes for each validated survey tool. If means are greater than 4, then the study is considered acceptable, appropriate, and/or feasible.
Time Frame: post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  Acceptability of Intervention Measure (AIM) | 4.5 (0.7)
  Intervention Appropriateness Measure (IAM) | 4.5 (0.8)
  Feasibility of Intervention Measure (FIM) | 4.6 (0.5)

3. Secondary Outcome: Resilience
Description: Connor-Davidson Resilience scale (CD-RISC; scored 0-40, higher scores indicate greater resilience)
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 28.5 (7.0)
  post-PRISM | 31.8 (5.6)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0089, Paired t-Test; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [0.9 to 5.8], Standard Deviation 6.9

4. Secondary Outcome: Overall Post-Traumatic Growth Inventory
Description: Post-Traumatic Growth Inventory (PTGI; scored 0-105 with factor subscales ranging from 0-10 to 0-35; higher scores indicate more positive transformation). Sub-scores are summed together to receive the overall score.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 57.4 (28.7)
  post-PRISM | 67.8 (28.6)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0169, Paired t-Test; Mean Difference (Final Values) = 10.4, 95% CI 2-sided [2 to 18.8], Standard Deviation 23.8

5. Secondary Outcome: Post-Traumatic Growth Inventory: Personal Strength Sub-scale
Description: Post-Traumatic Growth Inventory (PTGI; scored 0-105; higher scores indicate more positive transformation). The Post-Traumatic Growth Inventory Personal Strength sub-scale is scored from 0-20 with higher scores indicating increased resilience, self-reliance, confidence, humility, etc.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 10.9 (6.0)
  post-PRISM | 13.2 (6.1)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0162, Paired t-Test; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [0.5 to 4.3], Standard Deviation 5.3

6. Secondary Outcome: Post-Traumatic Growth Inventory: New Possibilities Sub-scale
Description: Post-Traumatic Growth Inventory (PTGI; scored 0-105; higher scores indicate more positive transformation). The Post-Traumatic Growth Inventory New Possibilities sub-scale is scored from 0-25 with higher scores indicating an increase in new interests, perspectives, more adaptability and openness to new opportunities.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 11 (6.9)
  post-PRISM | 14.5 (7.1)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0144, Paired t-Test; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [0.7 to 6.1], Standard Deviation 7.6

7. Secondary Outcome: Post-Traumatic Growth Inventory: Improved Relationships Sub-scale
Description: Post-Traumatic Growth Inventory (PTGI; scored 0-105; higher scores indicate more positive transformation). The Post-Traumatic Growth Inventory Improved Relationship sub-scale is scored from 0-35 with higher scores indicating an increased sense of belonging, emotional vulnerability, empathy, more supportive, and have an increased ability to form stronger bonds with others.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 20 (9.9)
  post-PRISM | 22.9 (9.2)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0264, Paired t-Test; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [0.4 to 5.5], Standard Deviation 7.3

8. Secondary Outcome: Post-Traumatic Growth Inventory: Spiritual Growth Sub-scale
Description: Post-Traumatic Growth Inventory (PTGI; scored 0-105; higher scores indicate more positive transformation). The Post-Traumatic Growth Inventory Spiritual Growth sub-scale is scored from 0-10 with higher scores indicating deeper and more meaningful beliefs, life philosophies and faith, more awareness, and a clearer purpose in life.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 6 (3.7)
  post-PRISM | 6.7 (3.7)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.1622, Paired t-Test; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.3 to 1.6], Standard Deviation 2.7

9. Secondary Outcome: Post-Traumatic Growth Inventory: Appreciation for Life Sub-scale
Description: Post-Traumatic Growth Inventory (PTGI; scored 0-105; higher scores indicate more positive transformation). The Post-Traumatic Growth Inventory Appreciation for Life sub-scale is scored from 0-15 with higher scores indicating increased gratitude, appreciation for the positive things in life, and clearer sense of priorities.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Out of 43 participants, only 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 9.5 (4.8)
  post-PRISM | 10.5 (4.7)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.1506, Paired t-Test; Mean Difference (Final Values) = 1, 95% CI 2-sided [-0.4 to 2.5], Standard Deviation 4

10. Secondary Outcome: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being
Description: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being tool (FACIT-Sp; scored 0-48 with each factor scored 0-16, higher scores indicate greater spiritual well-being). The overall score is a summation of each sub-score.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 37.1 (8.2)
  post-PRISM | 40.5 (5.4)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0012, Paired t-Test; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [1.5 to 5.4], Standard Deviation 5.5

11. Secondary Outcome: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being: Meaning Sub-score
Description: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being tool (FACIT-Sp; scored 0-48 with higher scores indicate greater spiritual well-being). The Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Meaning sub-scale is scored from 0-16 with one question reverse coded. Item scores for the sub-scale are summed, multiplied by 4, and divided by the number of items answered by the participant. A higher score indicates a greater sense of a meaningful life.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 13.2 (3)
  post-PRISM | 14.5 (1.7)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0021, Paired t-Test; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.5 to 2], Standard Deviation 2.1

12. Secondary Outcome: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being: Peace Sub-score
Description: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being tool (FACIT-Sp; scored 0-48 with higher scores indicate greater spiritual well-being). The Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Peace sub-scale is scored from 0-16 with one question reverse coded. Item scores for the sub-scale are summed, multiplied by 4, and divided by the number of items answered by the participant. A higher score indicates a greater sense of inner peace or harmony.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 11 (3.4)
  post-PRISM | 12.5 (2.6)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0027, Paired t-Test; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.6 to 2.4], Standard Deviation 2.6

13. Secondary Outcome: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being: Faith Sub-score
Description: Functional Assessment of Chronic Illness Therapy Spiritual Well-Being tool (FACIT-Sp; scored 0-48 with higher scores indicate greater spiritual well-being). The Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Faith sub-scale is scored from 0-16. Item scores for the sub-scale are summed, multiplied by 4, and divided by the number of items answered by the participant. A higher score indicates a greater sense of faith and spiritual beliefs.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 12.9 (3.7)
  post-PRISM | 13.6 (2.9)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0494, Paired t-Test; Mean Difference (Final Values) = 0.6970, 95% CI 2-sided [0.0 to 1.4], Standard Deviation 2

14. Secondary Outcome: Patient Activation Measure
Description: Patient Activation Measure (PAM; scored 0-100, higher scores indicate greater activation)
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 41.3 (5.4)
  post-PRISM | 41.9 (5.2)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.4707, Paired t-Test; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.1 to 2.3], Standard Deviation 4.8

15. Secondary Outcome: Fear of Cancer Recurrence Inventory
Description: Fear of Cancer Recurrence Inventory (FCRI-SF; scored 0-36, higher scores indicate greater fear of cancer recurrence)
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 17.9 (7.1)
  post-PRISM | 15.4 (7.1)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0082, Paired t-Test; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-4.3 to -0.7], Standard Deviation 5.1

16. Secondary Outcome: Patient Health Questionnaire
Description: Patient Health Questionnaire (PHQ-8; scored 0-24, higher scores indicate worse depressive symptoms)
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 6.4 (5.4)
  post-PRISM | 5.2 (4.3)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.1327, Paired t-Test; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.7 to 0.4], Standard Deviation 4.3

17. Secondary Outcome: General Anxiety Disorder Anxiety Scale
Description: General Anxiety Disorder Anxiety Scale (GAD-7; scored 0-21, higher scores indicate worse anxiety)
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
Scores on a scale
  pre-PRISM | 6.2 (5.8)
  post-PRISM | 5.1 (4.4)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.2046, Paired t-Test; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.9 to 0.6], Standard Deviation 5

18. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Global Health: Physical Health
Description: Patient-Reported Outcomes Measurement Information System Global Health - Physical Health (PROMIS-Global; physical health scored 4-20 with T-scores ranging from 16.2-67.7 and standard errors ranging from 4.8-5.9). A T-score of 50 represents the mean for the general population with a standard deviation of 10. A higher T-score indicates better physical health. A lower T-score would indicate a decrease in physical health.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
T-score
  pre-PRISM | 44.7 (9.1)
  post-PRISM | 44 (8.6)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.5252, Paired t-Test; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.8 to 1.4], Standard Deviation 5.9

19. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Global Health: Mental Health
Description: Patient-Reported Outcomes Measurement Information System Global Health - Mental Health (PROMIS-Global; mental health scored 4-20 with T-scores ranging from 21.2-67.6 and standard errors ranging from 4.6-5.3). A T-score of 50 represents the mean for the general population with a standard deviation of 10. A higher T-score indicates better mental health. A lower T-score would indicate a decrease in mental health.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Of 43 participants, 33 completed both surveys to obtain a pre/post value for each measure.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 33
T-score
  pre-PRISM | 45.7 (8.3)
  post-PRISM | 46.5 (8.8)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.4569, Paired t-Test; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.3 to 2.9], Standard Deviation 6

20. Secondary Outcome: Cholesterol
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: Biomarkers were only collected on participants with early-stage breast cancer (n=32). Of the 32 participants, 25 completed both surveys, biomarker collection timepoints, and all PRISM sessions.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
mg/dL
  pre-PRISM | 184.8 (33.3)
  post-PRISM | 196.9 (53.4)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.1497, Paired t-Test; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [-4.7 to 29.0], Standard Deviation 40.8

21. Secondary Outcome: Triglycerides
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
mg/dL
  pre-PRISM | 123.4 (80.4)
  post-PRISM | 140 (97.1)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.2163, Paired t-Test; Mean Difference (Final Values) = 16.6, 95% CI 2-sided [-10.4 to 43.7], Standard Deviation 65.5

22. Secondary Outcome: High Density Lipoprotein
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
mg/dL
  pre-PRISM | 52.7 (14.5)
  post-PRISM | 56.3 (15.6)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.0915, Paired t-Test; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-0.6 to 7.7], Standard Deviation 10.1

23. Secondary Outcome: Low Density Lipoprotein
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
mg/dL
  pre-PRISM | 107.4 (26.1)
  post-PRISM | 112.6 (41.4)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.3573, Paired t-Test; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-6.3 to 16.9], Standard Deviation 28.1

24. Secondary Outcome: Urea
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
mg/dL
  pre-PRISM | 14.7 (4.6)
  post-PRISM | 13.9 (5.9)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.3741, Paired t-Test; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.8 to 1.1], Standard Deviation 4.7

25. Secondary Outcome: Albumin
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
g/dL
  pre-PRISM | 4.2 (0.3)
  post-PRISM | 4.3 (0.2)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.6187, Paired t-Test; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.6 to 1.0], Standard Deviation 0.4

26. Secondary Outcome: Creatinine
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
mg/dL
  pre-PRISM | 1.1 (0.3)
  post-PRISM | 1.2 (0.4)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.3572, Paired t-Test; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.04 to 0.1], Standard Deviation 0.2

27. Secondary Outcome: Serum Cortisol
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
mg/dL
  pre-PRISM | 7.7 (4.3)
  post-PRISM | 9.6 (5.3)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.1080, Paired t-Test; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-0.5 to 4.3], Standard Deviation 5.8

28. Secondary Outcome: Homocysteine
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
umol/L
  pre-PRISM | 8.5 (3.7)
  post-PRISM | 9.5 (4.7)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.2088, Paired t-Test; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.6 to 2.5], Standard Deviation 3.7

29. Secondary Outcome: HbA1c
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
Participants
  pre-PRISM: Normal (<5.7%) | 9
  pre-PRISM: Pre-diabetic (5.7-6.4%) | 13
  pre-PRISM: Diabetic (>6.4%) | 3
  post-PRISM: Normal (<5.7%) | 11
  post-PRISM: Pre-diabetic (5.7-6.4%) | 9
  post-PRISM: Diabetic (>6.4%) | 5

30. Secondary Outcome: C-Reactive Protein
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
Participants
  pre-PRISM: Low Risk (<1 mg/L) | 2
  pre-PRISM: Average Risk (1-3 mg/L) | 10
  pre-PRISM: High Risk (>3 mg/L) | 13
  post-PRISM: Low Risk (<1 mg/L) | 2
  post-PRISM: Average Risk (1-3 mg/L) | 10
  post-PRISM: High Risk (>3 mg/L) | 13

31. Secondary Outcome: Tumor Necrosis Factor Alpha
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
pg/mL
  pre-PRISM | 1.4 (0.6)
  post-PRISM | 1.4 (0.5)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.7333, Paired t-Test; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.1 to 0.2], Standard Deviation 0.4

32. Secondary Outcome: Interleukin-6
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
pg/mL
  pre-PRISM | 1.7 (1.9)
  post-PRISM | 1.9 (2.3)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.6382, Paired t-Test; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.8 to 1.3], Standard Deviation 2.5

33. Secondary Outcome: Allostatic Load
Description: One point was assigned if BMI>30, systolic (SBP)>140 mmHg or diastolic blood pressure (DBP)>90 abstracted from the closest clinical encounter to the baseline visit, high-sensitivity C-reactive protein >0.41 mg/dL, HgbA1c>5.4, albumin<4 gm/dL and/or creatinine clearance <59 ml/min, total cholesterol >240 and/or triglycerides >150 mg/dL. The score range for this measure ranged from 0-9 with higher scores indicating a higher burden of stress or strain on the patient's body that can lead to worse outcomes.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
Scores on a scale
  pre-PRISM | 3.9 (1.4)
  post-PRISM | 3.7 (1.7)
Statistical Analysis 1: Comparison: PRISM Intervention; Test type: Other — Single group; p = 0.4771, Paired t-Test; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.8 to 0.4], Standard Deviation 1.4

34. Secondary Outcome: Nail Cortisol
Description: Biomarker samples were taken prior to and approximately one month after the last PRISM intervention session.
Time Frame: pre-PRISM (Baseline) and post-PRISM (ranged from 1 to 7 months after baseline)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention
Number analyzed (Participants) | 25
Participants
  pre-PRISM: Low (<=0.125) | 14
  pre-PRISM: Moderate (0.126-0.724) | 3
  pre-PRISM: High (>=0.725) | 6
  pre-PRISM: unknown | 2
  post-PRISM: Low (<=0.125) | 4
  post-PRISM: Moderate (0.126-0.724) | 10
  post-PRISM: High (>=0.725) | 4
  post-PRISM: unknown | 7

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | PRISM Intervention
All-Cause Mortality (participants affected / at risk) | 3/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

LIMITATIONS AND CAVEATS:
This pilot has several limitations as this was an initial feasibility study. The sample size was small and collected from a single site, there was not a control comparison, and the outcomes focused on feasibility. Thus, our study was not designed to evaluate efficacy. Additionally, sample heterogeneity could influence participants' psychological experiences while receiving PRISM intervention, and the sample size of this study did not permit sub-group analyses to address these differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT06133348/Prot_SAP_000.pdf